CLINICAL TRIAL: NCT00003172
Title: Randomized Phase II Trial of Either 5-Fluorouracil, Recombinant Alfa-2a-Interferon and Intravenous Hydroxyurea With Filgrastim Support (FHIG) or Doxorubicin/Docetaxel (Dd) in Patients With Advanced Gastric Cancer
Brief Title: Comparison of Combination Chemotherapy Regimens in Treating Patients With Advanced Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065978; E-6296
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2002-09

CONDITIONS: Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Filgrastim; Interferon-alpha; Docetaxel; Doxorubicin; Fluorouracil; Hydroxyurea

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: hydroxyurea

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different combinations and combining them with interferon alfa and G-CSF may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of different combination chemotherapy regimens in treating patients with advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the objective response rates for two different regimens in patients with advanced gastric cancer: the combination of fluorouracil plus hydroxyurea given as high dose 24 hour infusions plus interferon alfa-2a and filgrastim; versus the combination of doxorubicin and docetaxel. II. Evaluate the toxicities and reversibility of toxicities of each of these combinations in patients with advanced gastric cancer.

OUTLINE: This is an open label, two arm, multicenter, randomized study. Arm I: Patients receive fluorouracil (5-FU), recombinant alfa-2a interferon, hydroxyurea (HU), and filgrastim (granulocyte colony-stimulating factor; G-CSF). 5-FU is administered by 24 hour infusion on days 1, 8, 15, 22, 29, and 36 (weeks 1-6). Recombinant alfa-2a interferon is administered subcutaneously immediately before beginning the 5-FU infusion, then three times a week for 6 weeks. HU is administered by 24 hour infusion on days 1, 8, 15, 22, 29, and 36 (weeks 1-6). G-CSF is administered subcutaneously on days 3, 4, 5, and 6 on weeks 1-6. Weeks 7 and 8 are rest periods. Arm II: Patients receive doxorubicin administered by slow IV push followed (30 minutes after infusion) by docetaxel as a 1 hour IV infusion. Treatment is repeated every 21 days. All patients are assessed monthly during study and continue study treatment as long as no disease progression or unacceptable toxic effects are observed. Patients are followed every 3 months for the first 2 years, then every 6 months for years 2-5, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 26 patients (13 in each arm) and a maximum of 80 patients (40 in each arm) will be accrued in this study in approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction beyond the scope of surgical resection Must have measurable disease in either one or two dimensions either radiographically or by physical examination Measurable disease must be documented outside of a prior radiation portal Evaluable disease only not allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC greater than 4,000/mm3 Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT no greater than 1.5 times ULN Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease No chronic or unstable angina No uncontrolled congestive heart failure No arrhythmia No chronic angina No myocardial infarction in the past 1 year If history of atherosclerotic heart disease, prior cardiac catheterization or thallium stress test must not suggest coronary artery disease Neurology: No symptomatic peripheral neuropathy greater than grade 2 No cerebellar disease No seizure disorder No organic mental syndrome No major psychoaffective disorder Pulmonary: No chronic obstructive pulmonary disease No chronic bronchitis, emphysema, sarcoid, or bronchiectasis Other: No poorly controlled diabetes mellitus No psychiatric illness No active infections, including AIDS, ARC, or HIV positive No history of hypersensitivity to products containing Polysorbate 80 No history of uncontrolled alcohol or drug abuse No uncontrolled hypercalcemia No other prior malignancy within the past 5 years other than nonmelanomatous skin cancer or cervical carcinoma in situ Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior systemic chemotherapy Endocrine therapy: No chronic use of steroids No concurrent hormonal therapy (except birth control pills) Radiotherapy: At least 1 month since prior radiotherapy No concurrent palliative radiotherapy (arm I patients) Surgery: Must have fully recovered from surgery Other: At least 4 weeks since other investigational agents and recovered from all toxic effects No chronic use of aspirin, nonsteroidal antiinflammatory agents, antianginal medications, or extraordinary antihypertensive regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-12; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wadler, MD, Study Chair — Albert Einstein College of Medicine
Locations (25):
- United States (24):
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Wadler S, Brain C, Catalano P, Einzig AI, Cella D, Benson AB 3rd. Randomized phase II trial of either fluorouracil, parenteral hydroxyurea, interferon-alpha-2a, and filgrastim or doxorubicin/docetaxel in patients with advanced gastric cancer with quality-of-life assessment: eastern cooperative oncology group study E6296. Cancer J. 2002 May-Jun;8(3):282-6. doi: 10.1097/00130404-200205000-00013. PMID 12074329
- [Result] Wadler S, Einzig A, Catalano P, et al.: Randomized phase II trial of either flourouracil (F), parenteral hydroxyurea (H), interferon-alfa-2a (I) and filgrastim (G) or doxorubicin/docetaxel (AD) in patients (PTS) with advanced gastric cancer: Eastern Cooperative Oncology Group (ECOG) study EST 6296. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-659, 2001.